CLINICAL TRIAL: NCT05378295
Title: Personalized Microbial Substrates to Prevent Type 2 Diabetes
Brief Title: Personalized Fiber and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL76905.068.21
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isocaloric fermentable oligosaccaride (Active Comparator): isocaloric fermentable oligosaccaride
  Interventions: Dietary Supplement: Fermentable oligosaccharide
- Personalized fiber mixture (Experimental): 12 g for 2 weeks, followed by 24 g for 10 weeks
  Interventions: Dietary Supplement: Personalized fiber mixture

INTERVENTIONS:
Dietary Supplement: Fermentable oligosaccharide — Supplementation period 12 weeks
  Arms: isocaloric fermentable oligosaccaride
Dietary Supplement: Personalized fiber mixture — Supplementation period 12 weeks
  Arms: Personalized fiber mixture

SUMMARY:
In this project the investigators intend to study the therapeutic potential of a personalized fibre mixture in individuals at high risk of developing T2DM, and aim to address the following key objectives:

1. To investigate whether a mixture of fermentable fibres, which differ in DP and side chains, will stimulate a broad range of SCFA-producing bacterial genera, resulting in enhanced chronic SCFA production throughout the whole colon with a large variation between individuals;
2. To unravel whether providing personalized fibre mixtures, selected based on the individuals' initial microbiota and capacity for SCFA production is crucial to successfully improve host insulin sensitivity and metabolic health

ELIGIBILITY:
Inclusion Criteria:

Overweight/obese insulin resistant/prediabetic participants (age 30-70 y, BMI ≥ 28 kg/m2 < 40 kg/m2)

Exclusion Criteria:

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥ 7.0 mmol/L and 2h glucose ≥ 11.1 mmol/L)
* Gastroenterological diseases or abdominal surgery;
* Cardiovascular diseases, cancer, liver or kidney malfunction, disease with a life expectancy shorter than 5 years;
* Abuse of products; alcohol and drugs, excessive nicotine use defined as >20 cigarettes per day;
* Plans to lose weight or following of a hypocaloric diet;
* Regular supplementation of pre- or probiotic products, use of pre- or probiotics 3 months prior to the start of the study;
* Intensive exercise training more than three hours a week;
* Use of any medication that influences glucose or fat metabolism and inflammation (i.e. NSAIDs);
* Regular use of laxation products;
* Use of antibiotics in the last three months (antibiotics use can alter substantially the gut microbiota composition).
* Follow a vegetarian diet.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Peripheral insulin sensitivity | Before and 12 week after the start of the intervention
  The change of peripheral insulin sensitivity (m-value) as assessed by a hyperinsulinaemic-euglycemic clamp

SECONDARY OUTCOMES:
Energy expenditure (indirect calorimetry) | Before and 12 week after the start of the intervention
  The change in energy expenditure as measured via ventilated hood system
Substrate oxidation (indirect calorimetry) | Before and 12 week after the start of the intervention
  The change in substrate oxidation as measured via ventilated hood system
circulating SCFA | Before and 12 week after the start of the intervention
  The change in concentrations of circulating SCFA
Faecal SCFA | Before and 12 week after the start of the intervention
  The change in concentrations of faecal SCFA
Faecal microbiota composition and in vitro microbial activity testing | Before and 12 week after the start of the intervention
  The change in faecal microbiota composition assessing abundances of bacteria and diversity indices as assessed via 16s rRNA gene
Circulating hormones such as insulin | Before and 12 week after the start of the intervention
  The change in concentrations of circulating hormones in peripheral blood
Circulating metabolites such as glucose | Before and 12 week after the start of the intervention
  The change in concentrations of metabolites in peripheral blood
body fat percentage | Before and 12 week after the start of the intervention
  The change in body fat percentage as assessed using DEXA scans
fat mass | Before and 12 week after the start of the intervention
  The change in fat mass in kg as assessed using DEXA scans
lean mass | Before and 12 week after the start of the intervention
  The change in lean mass in kg as assessed using DEXA scans
visceral fat | Before and 12 week after the start of the intervention
  The change in visceral fat in gram as assessed using DEXA scans
body weight | Before and 12 week after the start of the intervention
  The change in body weight in kg using a weight scale

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided